CLINICAL TRIAL: NCT07298343
Title: A Phase II, Double-blind, Randomised, Placebo-controlled Trial to Evaluate the Efficacy and Tolerability of ZED1227 in Celiac Disease Subjects Experiencing Symptoms Despite Gluten-free Diet
Brief Title: Evaluating the Efficacy and Tolerability of ZED1227 in Subjects With Non-responsive Celiac Disease
Acronym: CEC-013/CEL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEC-013/CEL; 2023-506150-21 (EudraCT Number)
Record Dates: First submitted 2025-12-17; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Celiac Disease
Keywords: Celiac Disease; non-responsive Celiac Disease
MeSH Terms: conditions — Celiac Disease | interventions — ZED1227

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- low Dose 1 ZED1227 + SIGE (Experimental)
  Interventions: Drug: ZED1227 + SIGE
- Placebo + SIGE (Placebo Comparator)
  Interventions: Other: Placebo
- medium Dose ZED1227 + SIGE (Experimental)
  Interventions: Drug: ZED1227 + SIGE
- high dose ZED1227 + SIGE (Experimental)
  Interventions: Drug: ZED1227 + SIGE
- low Dose 2 ZED1227 + SIGE (Experimental)
  Interventions: Drug: ZED1227 + SIGE

INTERVENTIONS:
Drug: ZED1227 + SIGE — oral treatment with different daily doses of ZED1227 vs placebo
  Arms: high dose ZED1227 + SIGE; low Dose 1 ZED1227 + SIGE; low Dose 2 ZED1227 + SIGE; medium Dose ZED1227 + SIGE
Other: Placebo — Placebo + SIGE
  Arms: Placebo + SIGE

SUMMARY:
A study to discover if ZED1227 can improve continued celiac disease symptoms despite a gluten-free diet

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Men or women between 18 and 80 years of age, inclusively
* Documented initial biopsy-proven diagnosis of celiac disease or, in case of missing histological documentation, TG2-IgA > 10 x upper limit of normal (ULN) at diagnosis at least 12 months prior to V0
* Adherence to a gluten-free diet (GFD) for at least 12 months prior to V0
* Human leukocyte antigen DQ (HLA-DQ) typing compatible with celiac disease

Exclusion Criteria:

* Presence of hypo- or hyperthyroidism. A patient with a well-controlled thyroid disorder during the previous 3 months can be included
* Patients diagnosed to have confirmed refractory celiac disease type I (RCDI) or II (RCDII), with the exception that patients with a diagnosis of RCDI can be considered for inclusion if they do not have clear signs of T cell monoclonality or atypical T cells (e.g., as revealed by CD3/CD8 immunohistochemistry) and if they do not present with very severe symptoms and/or parameters of significant malabsorption and if they have not received prior treatment with immunosuppressants such as budesonide or azathioprine,
* Severe complications of celiac disease
* Concomitant diseases of the intestinal tract in addition to celiac disease, such as Crohn's disease, ulcerative colitis, other forms of inflammatory bowel disease, severe irritable bowel syndrome, microscopic colitis, small intestinal bacterial overgrowth (SIBO), exocrine pancreatic insufficiency; any other active diseases of the intestinal tract (e.g., active, untreated peptic ulcer, esophagitis, gastroesophageal reflux disease) that might, in the investigator's opinion, interfere with assessment of symptoms of abdominal pain, diarrhoea, or other components of celiac disease
* History or presence of dermatitis herpetiformis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in CDSD GI Specific Symptom Score | 12 weeks

SECONDARY OUTCOMES:
Change in PRO: Change from baseline in the percentage of Symptom Free Days (SFD) | V5 (Wk 15) over a 14-day period
Histological assessment of villous height to crypt depth ratio (VH:CrD) | 15 weeks
Change in CDSD Non-Stool GI Symptom Score (abdominal pain, bloating, nausea) | 12 weeks
Proportion of subjects with histologic non-worsening, defined as change in VH:CrD ≥ 0 | 15 weeks
Change in duodenal mucosal inflammation measured as the density of CD3positive intraepithelial lymphocytes (IELs) | 15 weeks
Change in serological markers TG2-IgA, TG2-IgG, DGP-IgA, DGP-IgG, and EmA-IgA | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Mainz, Mainz, Germany

IPD SHARING:
Plan to Share IPD: No